CLINICAL TRIAL: NCT04505735
Title: Amyloid Imaging With 11C-PiB in Healthy Aging and Mild Cognitive Impairment
Status: Terminated | Type: Observational
Why Stopped: Issues with local production of 11-cPiB radiotracer
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2064
Record Dates: First submitted 2020-07-29; First posted 2020-08-10 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Alzheimer Disease; Healthy Aging
Keywords: Healthy Older Adults; Mild Cognitve Impairment; Imaging; C-PiB
MeSH Terms: conditions — Alzheimer Disease | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Control: Adults with no history of memory complaints, diagnosis of MCI, or dementia from a physician
  Interventions: Drug: 11C-PiB
- Adults with Mild Cognitive Impairment: Adults with cognitive decline verified by a study partner or cognitive impairment verified by the study physician. The cognitive decline has had limited impact on functional activities; general cognition and functional performance are sufficiently preserved such that a diagnosis of dementia cannot be made by the enrolling physician
  Interventions: Drug: 11C-PiB

INTERVENTIONS:
Drug: 11C-PiB — Pittsburgh Compound-B (11C-PiB) is a diagnostic imaging agent that binds to beta-amyloid plaques and allows them to be viewed using positron emission tomography (PET) imaging.
  Other Names: Pittsburgh compound B

SUMMARY:
The purpose of this study is to measure the amount of amyloid in the brain. Amyloid is a protein found in the brain of patients with Alzheimer's disease and can be detected using a Positron Emission Tomography (PET) scan. This study is interested in how amyloid levels in the brain relate to memory and thinking abilities.

DETAILED DESCRIPTION:
The overarching goal of this study is to use 11C-PiB, a commonly used tracer that binds to amyloid plaques in the brain, as a biological marker of Alzheimer's disease (AD) related brain changes. Data from this PET-only study will be compared to and analyzed with data from the Investigators' longitudinal biomarker studies, COMIRB #15-1774 and COMIRB #18-2607. This enables investigators to examine how deposition of the amyloid protein relates to cognitive aging in both symptomatic and asymptomatic older adults. It will assist investigators in comparing rates of change in memory and thinking ability in healthy subjects who are amyloid positive versus amyloid negative, as well as in comparing rates of conversion to a higher level of impairment (e.g. such as Mild Cognitive Impairment converting to Alzheimer's Disease) based on the quantitative analysis of amyloid burden. Moreover, by capitalizing on data across the two studies, the investigators will be able to better understand the relationship between amyloid deposition (as assessed by PET; current proposal) and other biomarkers (as assessed in COMIRB #15-1774, COMIRB #18-2607), which ultimately may help the investigators better predict the onset and progression of clinical AD symptoms. Participants will be recruited solely from the longitudinal study (COMIRB # 15-1774) in order to provide data comparison on an individual and group basis.

The goals of this study are as follows:

1. Evaluate the relationship between amyloid burden, as assessed by 11C-PiB, with both cross-sectional and longitudinal biomarkers (e.g. blood; nasal biopsy; CSF; MRI; DNA) obtained in the longitudinal study (COMIRB # 15-1774, COMIRB #18-2607).
2. Compare rates of change in memory and other cognitive abilities (obtained in COMIRB # 15-1774, COMIRB #18-2607) in healthy subjects who show elevated amyloid deposition with those who are "amyloid negative".
3. Evaluate the relationship between amyloid burden and health history, informant report of subjective cognitive and psychiatric difficulties, and participant-reported psychiatric symptoms.
4. Investigate predictive utility of amyloid burden in identifying individuals most at risk for conversion (e.g. healthy controls to MCI, and MCI to AD).
5. Identify why a subset of "amyloid positive" individuals do not show symptoms of clinical AD or delay conversion to MCI or AD.

ELIGIBILITY:
Inclusion Criteria:

Patients may be enrolled in the Normal Control group if the following criteria are met:

1. Males or nonpregnant females ≥ 50 years of age;
2. Have no history of memory complaints;
3. Have no diagnosis of MCI or dementia from a physician
4. Currently enrolled in the Rocky Mountain Alzheimer's Disease Center at the University of Colorado School of Medicine (RMADC at UCSOM) Longitudinal Biomarker and Clinical Phenotyping Study (COMIRB #15-1774) or Longitudinal Innate Immunity and Aging study (LIIA; COMIRB #18-2607)
5. Willing to have clinical research information from the Longitudinal Biomarker and Clinical Phenotyping Study (COMIRB #15-1774) and/or LIIA (COMIRB #18-2607) study shared/combined with the current study.
6. Participated in the MRI procedure for COMIRB #15-1774 or COMIRB #18-2607.

Patients may be enrolled in the Mild Cognitive Impairment (not demented) group if the following criteria are met:

1. Males or nonpregnant females ≥ 50 years of age;
2. Have cognitive decline verified by a study partner or cognitive impairment verified by the study physician. The cognitive decline has had limited impact on functional activities; general cognition and functional performance are sufficiently preserved such that a diagnosis of dementia cannot be made by the enrolling physician
3. Have a Clinical Dementia Rating score of 0.5*
4. Can tolerate a 70-minute PET scan. The Principal Investigator and Co-PI will carefully assess each patient and use sound judgment to determine whether the patient can tolerate the PET scan procedure;
5. Ability to provide informed consent for study procedures (If the patient is ineligible to give informed consent, based on local standards, the patient's legally authorized representative may consent on behalf of the patient but the patient must still confirm assent. This person may serve as the study partner as well).
6. Concurrently enrolled in the Rocky Mountain Alzheimer's Disease Center at the University of Colorado School of Medicine (RMADC at UCSOM) Longitudinal Biomarker and Clinical Phenotyping Study (Bio-AD; COMIRB #15-1774) or Longitudinal Innate Immunity and Aging study (LIIA; COMIRB #18-2607)
7. Participated in the MRI procedure for COMIRB #15-1774 or COMIRB #18-2607.
8. Willing to have clinical research information from the Longitudinal Biomarker and Clinical Phenotyping Study (COMIRB #15-1774) and/or LIIA (COMIRB #18-2607) study shared/combined with the current study.

   * For aging adults with atypical phenotypes (e.g., early onset Alzheimer's Disease; Posterior Cortical Atrophy; Logopenic variant primary progressive aphasia), a CDR of 1 will be accepted if the study team determines that their severity is mild. The reason for this caveat is that these phenotypes often reach a CDR of 1 quickly due to cortical symptoms (e.g., loss of visual perception); in these cases, the CDR may overestimate their true severity level.

Exclusion Criteria:

Patients will be excluded from enrollment if they:

1. Have a current serious or unstable illness that in the enrolling physician's opinion, could interfere with completion of the safety or efficacy evaluations included in this study.
2. Have a known brain lesion, pathology or alternative diagnosis that strongly explains the patient's clinical presentation;
3. Are receiving any investigational medications, or have participated in a trial with investigational medications within the last 30 days;
4. Have had a clinical radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session; have had a research radiopharmaceutical imaging study done within 12 months or have one planned in the next 12 months.
5. Exposed to radiation in the work place during the previous year

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Rocky Mountain Alzheimer's Disease Center at the University of Colorado School of Medicine (RMADC at UCSOM) Longitudinal Biomarker and Clinical Phenotyping Study (Bio-AD; COMIRB #15-1774) and/or Longitudinal Innate Immunity and Aging study (LIIA; COMIRB #18-2607).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Amyloid burden | Single visit PET scan (Day 0)
  Amyloid burden will be calculated using the standardized uptake volume ratio (SUVr) to do a centiloid analysis. This is assessed on a 100-point scale, the "Centiloid" (CL), where the data is scaled so that an average value of zero is amyloid-negative subjects and an average value of 100 is a typical Alzheimer's Disease patient (with negative numbers and numbers above 100 being possible). The site will scale the data along this 0-100 scale to determine amyloid burden in relation to Alzheimer's disease and compare to data from COMIRB #15-1774 or COMIRB #18-2607

CONTACTS AND LOCATIONS:
Overall Officials: Brianne M Bettcher, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No